CLINICAL TRIAL: NCT05341141
Title: Effectiveness of Cryotherapy Combined With Compression Therapy in Preventing Albumin-paclitaxel Induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: Effectiveness of Cryotherapy Combined With Compression Therapy for Preventing Chemotherapy-induced Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-P30(FZQ)
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: Chemotherapy-induced Peripheral Neuropathy; Albumin-paclitaxel; Cryotherapy; Compression Therapy; dose-dense chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ddEC-ddT and cryotherapy combined with compression (Experimental): Cryotherapy will be applied using a frozen glove and sock for 15 minutes before, during and 15 minutes after each albumin-paclitaxel infusion. Compression therapy will be applied using a surgical glove for 30 minutes before, during and 30 minutes after each albumin-paclitaxel infusion.
  Interventions: Device: Frozen glove and sock; Drug: ddEC-ddT
- ddEC-ddT (Other): ddEC-ddT will be administered without cryotherapy combined with compression.
  Interventions: Drug: ddEC-ddT

INTERVENTIONS:
Device: Frozen glove and sock — Preparation of frozen glove and sock: 4℃ for 3 hours.
  Arms: ddEC-ddT and cryotherapy combined with compression
Drug: ddEC-ddT — Epirubicin (E) 90~100mg/m^2, i.v., d1 + cyclophosphamide (C) 600 mg/m^2, i.v., d1, q2w, for 4 cycles followed by albumin-paclitaxel (T) 260 mg/m^2, i.v., d1, q2w, for 4 cycles.
  Other Names: Chemotherapy

SUMMARY:
This is a prospective, multi-center, randomized study designed to evaluate the clinical efficacy of cryotherapy combined with compression therapy in preventing albumin-paclitaxel induced peripheral neuropathy.

DETAILED DESCRIPTION:
All HER-2 negative breast cancer patients received neoadjuvant chemotherapy with four cycles of dose-dense epirubicin and cyclophosphamide (ddEC) followed by four cycles of dose-dense albumin-paclitaxel (ddT). The patients were randomly assigned in a 1:1 ratio to receive cryotherapy combined with compression or no intervention. The primary endpoint was incidence of grade 3 and higher peripheral neuropathy as assessed by NCI-CTCAE V5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged from 20 to 70 years old;
2. Histologically confirmed as invasive breast cancer;
3. HER-2 negative (defined by IHC 0 or 1+ ,or FISH negative);
4. Participants who meet any of the following conditions: 1) T > 2 cm, ER<1% and PR<1%; 2) T > 2 cm, ER≥1% and biopsy pathology (FNAB or CNB) diagnosed regional lymph node metastasis;
5. Without any previous treatment;
6. ddEC-ddT neoadjuvant chemotherapy is planned;
7. Participants must have at least one measurable disease according to RECIST 1.1;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
9. LVEF ≥ 50%;
10. The ECG results are judged to be almost normal or normal, or the investigator judges that the abnormalities are not clinically significant;
11. Bone marrow function: absolute neutrophil counts (ANC) ≥ 1.5x10^9/L, platelets ≥ 100x10^9/L, hemoglobin ≥ 90g/L;
12. Liver and kidney function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are both ≤2.5 ULN; serum total bilirubin and serum creatinine are both ≤ 1.5 ULN;
13. Participants had good compliance with the planned treatment and follow-up, understood the study procedures of this study, and signed informed consent form.

Exclusion Criteria:

1. Breast cancer with distant metastasis;
2. A history of other malignancies;
3. In the past or present, participants with sensory or motor neurological diseases;
4. Participants who are known to be allergic to the active or other components of the study treatment;
5. Cerebral thrombosis is present;
6. In the past and present, participants with severe cardiac disease or discomfort , including but not limited: 1) High-risk uncontrolled arrhythmia, atrial tachycardia (heart rate > 100/min in resting state), significant ventricular arrhythmia (ventricular arrhythmia) or higher atrioventricular block (second-degree type 2 [Mobitz 2] atrioventricular block or third-degree atrioventricular block); 2) Angina pectoris requiring anti-angina medication; 3) Clinically significant valvular heart disease; 4) ECG showing transmural myocardial infarction; 5) ncontrolled hypertension (eg systolic blood pressure > 180mm Hg or diastolic blood pressure > 100mmHg); 6) Myocardial infarction; 7) Congestive heart failure;
7. Participants have the following serious illnesses or medical conditions, including but not limited: 1) History of serious neurological or psychiatric disorders, including psychosis, dementia, or epilepsy, that prevent understanding and informed consent; 2) Active uncontrolled infection; 3) Active pepticulcer, unstable diabetes;
8. Participants who are pregnant, breastfeeding, or refuse to use adequate contraception prior to study entry and for the duration of study participation;
9. Participants who were judged by the investigator to be unsuitable for this study.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 and higher peripheral neuropathy as assessed by NCI-CTCAE V5.0 | 4 years
  Incidence of grade 3 and higher peripheral neuropathy as assessed by NCI-CTCAE V5.0

SECONDARY OUTCOMES:
Incidence of grade 2 and higher peripheral neuropathy as assessed by NCI-CTCAE V5.0 | 4 years
  Incidence of grade 2 and higher peripheral neuropathy as assessed by NCI-CTCAE V5.0
Proportion of patients reporting level D and above based on the Patient Neurotoxicity Questionnaire (PNQ) | 4 years
  PNQ scale ranges from scores A to E; with scoring of A being not affected neuropathy, and E with the worst neuropathy.
EORTC QLQ-CIPN20 | 4 years
  The EORTC QLQ-CIPN20 is a fairly new 20-item questionnaire evaluating various aspects of CIPN. It has three subscales assessing sensory (nine items), motor (eight items), and autonomic (three items) symptoms and functioning with each item measured on an ordinal 1-4 scale (1, not at all; 4, very much).
Incidence and severity of other adverse events as assessed by NCI-CTCAE V5.0 | 4 years
  Incidence and severity of other adverse events as assessed by NCI-CTCAE V5.0
Total pathological complete response (tpCR) rate | Within 2 to 4 weeks after completion of neoadjuvant therapy
  Total pathological complete response (tpCR) was defined as the absence of invasive lesions in the breast and axillary lymph nodes (ypT0/is ypN0). The tpCR rate is the percentage of participants with tpCR.
Breast pathological complete response (bpCR) rate | Within 2 to 4 weeks after completion of neoadjuvant therapy
  Breast pathological complete response (bpCR) was defined as no invasive carcinoma in the breast (ypT0/is). The bpCR rate is the percentage of participants with bpCR.
Objective response rate (ORR) | After the last dose to before surgery or within 28 days
  The number of participants who achieved complete response and partial response at the end of neoadjuvant chemotherapy as a percentage of the overall evaluable participants.
Invasive disease-free survival (IDFS) | 3 years
  Invasive disease free survival was defined as the time from enrollment until the date of first occurrence of one of the following events: invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence (including first metastasis), invasive contralateral breast cancer, second primary invasive cancer (nonbreast, not including squamous or basal cell skin cancers, or new in situ carcinomas of any site), or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Fan, MD, Principal Investigator — Breast center at Peking University Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China